CLINICAL TRIAL: NCT06485739
Title: The Efficacy and Safety of Irinotecan Liposomes Combined With Cisplatin/Carboplatin for Gastrointestinal Pancreatic Neuroendocrine Carcinoma: a Real-world Study
Brief Title: Irinotecan Liposomes for the Treatment of Neuroendocrine Carcinoma
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, Li EnXiao, Medical professor, First Affiliated Hospital Xi'an Jiaotong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-101
Record Dates: First submitted 2024-06-27; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Neuroendocrine Tumors
Keywords: Irinotecan liposomes; Neuroendocrine tumors
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Irinotecan liposome combined administration group (Experimental): The combination of irinotecan liposomes and cisplatin or carboplatin regimen is recommended for treatment, with a recommended dose of 70mg/m2 for irinotecan liposomes. For UGT1A1 * 28 homozygous patients, the initial dose of irinotecan liposomes is adjusted to 50mg/m2. If the patient tolerates during the first treatment cycle, the dose can be adjusted to 70mg/m2 for subsequent treatment cycles; Every 4 weeks is a treatment cycle, with 6 cycles of treatment. If the researcher determines that the patient can continue to benefit from 6 cycles of treatment, the treatment will continue until 8 cycles;
  Interventions: Drug: Irinotecan liposomes combined with cisplatin/carboplatin

INTERVENTIONS:
Drug: Irinotecan liposomes combined with cisplatin/carboplatin — Irinotecan liposomes 70mg/m2，use on the first day of each cycle The dosage of cisplatin and carboplatin is determined by the researchers
  Other Names: Irinotecan liposomes group

SUMMARY:
This study is a real-world clinical study. It is expected to include 20 patients with first-line and second-line gastrointestinal pancreatic neuroendocrine carcinoma who will be treated with irinotecan liposomes combined with cisplatin or carboplatin regimen. The research unit is the First Affiliated Hospital of Xi'an Jiaotong University. The study includes a screening period (within 28 days), a treatment period (planned for 6 cycles), and a follow-up period (safety follow-up and PFS follow-up). The subjects signed an informed consent form and underwent baseline examination during the screening period. Patients who met the inclusion and exclusion criteria entered the treatment period. All subjects completed the relevant examinations specified in the protocol during the treatment process to observe safety, tolerance, and efficacy. The same subject only received one dosing plan during the study period. After the treatment period ends, enter the follow-up period.

DETAILED DESCRIPTION:
Neuroendocrine tumors (NENs) are a type of tumor originating from stem cells and possessing neuroendocrine markers that can produce bioactive amines and/or peptide hormones. Due to their heterogeneity and inertness, they have been defined as "carcinoids". Due to differences in origin, pathological grading, and treatment methods, NEN has different clinical manifestations and prognosis. Although NEN still meets the definition of rare disease, its incidence rate has increased significantly worldwide in the past decades. In the United States, the incidence rate of NEN in 2012 was 6.98/100000, about seven times the incidence rate reported in 1973 (1.09/100000). Among them, gastrointestinal and pancreatic neuroendocrine tumors (GEP NENs) are the most common type of NEN, accounting for 67.5% of all NEN cases. They mainly occur in the digestive tract or pancreas and can produce amine substances and peptide hormones such as glucagon, insulin, gastrin, or adrenocorticotropic hormone (ACTH).

We analyzed the data of ordinary irinotecan in first-line and second-line treatment of GEP-NEC and found that a prospective Phase II clinical study included 66 patients with advanced GEP-NEC. The results showed that the efficacy of the first line treatment using EP and IP regimens was equivalent, with an effective rate of over 40%. However, the efficacy of the second-line FOLFOX and FOLFIRI regimens is not ideal. Studies by HENTIC et al. have shown that the response rate of GEP-NEC to the FOLFIRI regimen is 31%, but the PFS is only 4 months; DU et al. also found that the median PFS of the FOLFIRI regimen was only 6.5 months in 11 patients with gastrointestinal NEC. The current research results on the FOLFOX regimen are similar. If there are studies showing that FOLFOX is used as a second-line regimen to treat 12 patients with advanced GEP-NEC, the median PFS is 4.5 months. HEETFELD et al. observed the efficacy of the FOLFIRI/FOLFOX regimen in GEP-NEC patients on the second or third line, and the results also showed a median PFS of 3.0 months and 2.5 months for the second and third line groups, respectively. Overall, the second-line treatment regimens recommended by the NCCN guidelines have not shown ideal efficacy and PFS in GEP-NEC.

Based on the literature review above and the birth of independently developed irinotecan liposomes by Shiyao, we plan to conduct a real-world study on the combination of irinotecan liposomes and platinum based treatment of gastrointestinal neuroendocrine carcinoma. The aim is to explore the efficacy and safety of a combination of irinotecan liposomes and platinum based chemotherapy regimen in first-line and second-line patients with gastrointestinal neuroendocrine carcinoma, providing better clinical evidence of efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* The patient fully understands this study, voluntarily participates and signs an informed consent form (ICF);
* Age: ≥ 18 years old;
* Expected survival time ≥ 3 months;
* Patients with high-grade gastrointestinal pancreatic neuroendocrine tumors (NET G3) and neuroendocrine cancers (NECs) confirmed by histopathology;
* Have not undergone or undergone a systematic anti-tumor treatment in the past;
* According to RECIST 1.1 standard, patients must have at least one measurable diameter target lesion (tumor lesion CT scan length ≥ 10mm, lymph node lesion CT scan short diameter ≥ 15mm, scan layer thickness 5mm);
* ECOG score 0-2 points;
* Absolute neutrophil count (ANC) ≥ 1.5 x 10 ^ 9/L, platelet count ≥ 100 x 10 ^ 9/L, and hemoglobin count ≥ 90 g/L;
* Liver and kidney function: serum creatinine ≤ 1.5 times the upper limit of normal value; AST and ALT ≤ 2.5 times the upper limit of normal values (≤ 5 times the upper limit of normal values for patients with liver invasion); Total bilirubin ≤ 1.5 times the upper limit of normal value (≤ 3 times the upper limit of normal value for patients with liver invasion);
* Women of childbearing age must undergo a pregnancy test (serum) within 7 days before enrollment, and the result is negative. They are willing to use appropriate methods of contraception during the trial period and 8 weeks after the last administration of the investigational drug;

Exclusion Criteria:

* Patients with neuroendocrine tumors G1 and G2;
* Has hypersensitivity to any investigational drug or its components;
* Diagnosed as intestinal obstruction through imaging;
* Uncontrollable systemic diseases (such as infection during the promotion period, uncontrollable hypertension, diabetes, etc.);
* Active infection of hepatitis B and hepatitis C (hepatitis B B virus surface antigen is positive and hepatitis B B virus DNA exceeds 1x103 copies/mL; hepatitis C virus RNA exceeds 1x103 copies/mL);
* Human Immunodeficiency Virus (HIV) infection (HIV antibody positive);
* Has previously or currently suffered from other malignant tumors (except for effectively controlled non melanoma skin basal cell carcinoma, breast/cervical carcinoma in situ, and other malignant tumors that have not been treated and have been effectively controlled within the past five years);
* Pregnant and lactating women, as well as patients of childbearing age who are unwilling to take contraceptive measures;
* Patients with other malignant tumors that require treatment;
* The researchers determined that patients who are not suitable to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Intracranial Objective response rate | Data obtained up until progression, or the last evaluable assessment in the absence of progression, will be assessed up to 1 years.
  Per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) using Investigator assessments, is defined as the number (%) of patients with tumour response of Complete Response or Partial Response, will be assessed up to 1 years.

SECONDARY OUTCOMES:
Complete Response | Data obtained up until progression, or the last evaluable assessment in the absence of progression, will be assessed up to 1 years.
  According to the solid tumor response evaluation criteria 1.1 (RECIST 1.1) evaluated by researchers, it is defined as the number of patients (%) whose target lesions disappear and whose short diameter of all pathological lymph nodes (including target and non target nodules) must be reduced to<10 mm, and will be evaluated within one year.
Progression-free survival | Progression-free survival (PFS) analysis based on investigator assessment per RECIST 1.1, and will be assessed up to 3 years.
  Progression-free survival (PFS) is defined as the time from first treatment recorded until the date of disease progression based on investigator assessment.
Overall Survival | The time from beginning of treatment until death due to any cause and will be assessed up to 3 years.
  Overall survival is defined as the time from beginning of treatment until death due to any cause and will be assessed up to 3 years.
Safety/Adverse event | From the recorded first dose of Furmonertinib to 4 weeks after the recorded last dose of Furmonertinib
  Incidence of Adverse Events (AEs): Incidence, severity and seriousness of adverse events, incidence of serious adverse events (SAEs), which usually be graded by CTCAE v5.0 based on current clinical practice.

CONTACTS AND LOCATIONS:
Overall Officials: EnXiao Li, PhD, Study Director — First Affiliated Hospital of Xian Jiaotong University

IPD SHARING:
Plan to Share IPD: No